CLINICAL TRIAL: NCT00813969
Title: A Phase I Study to Assess the Feasibility, Safety, and Tolerability of Autologous Mesenchymal Stem Cell Transplantation in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: Autologous Mesenchymal Stem Cell (MSC) Transplantation in MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-MSC-001
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Progressive Relapsing Multiple Sclerosis
Keywords: Mesenchymal Stem Cell; MSC; Autologous; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous MSC transplantation (Experimental)
  Interventions: Biological: Autologous mesenchymal stem cell transplantation

INTERVENTIONS:
Biological: Autologous mesenchymal stem cell transplantation — A single IV infusion of up to 2 million cells per kg based on the MSC numbers achieved after culture expansion

SUMMARY:
The study is an investigator-run, open-label Phase 1 safety study of autologous mesenchymal stem cell transplantation, involving approximately 24 ambulatory participants with relapsing forms of MS (approximately equal numbers with relapsing-remitting and secondary progressive/ progressive relapsing MS) and evidence of involvement of the anterior afferent visual system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55, inclusive.
* Diagnosis of MS
* Relapsing form of MS (relapsing-remitting, secondary progressive, or progressive-relapsing course).
* EDSS score 3.0-6.5, inclusive. (Must be able to walk)
* Active disease during prior 24 months.
* Documented evidence of involvement of the anterior afferent visual system: previous optic neuritis, optic atrophy or an afferent pupillary defect on exam, RNFL thickness on OCT <LLN in at least one eye OR documented VEP latency in at least 1 eye.
* Cranial MRI scan demonstrating T2-hyperintense lesions satisfying diagnostic criteria for MS
* Ability to perform the component tests of the MSFC (T25FW, 9HPT, PASAT3).
* Ability to perform SLCLA.
* Has given written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant infectious illness (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days of the Screening Visit.
* History of cancer other than basal cell carcinoma of the skin.
* History or laboratory results indicative of any significant cardiac, endocrine, hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, neoplastic, or other disorder that in the opinion of the Principal Investigator would preclude the safe performance of BM aspiration, infusion of autologous MSCs, or performance of any of the planned study assessments.
* Abnormal blood tests which exceed designated limits.
* Positive screening tests for hepatitis B, hepatitis C, HIV 1&2, HTLV I/II, CMV, West Nile virus, syphilis, blood parasite infection.
* Clinically significant abnormality on chest X-ray.
* Clinically significant abnormality on EKG.
* Oxygen-saturation <90% on room air.
* History of alcohol or drug abuse within one year.
* Any metallic material or electronic device in the body, or condition that precludes the participant from undergoing MRI with Gd administration.
* Uncontrolled glaucoma or other ocular condition that precludes performing OCT or interpreting the results.
* MS relapse with onset within 30 days prior to the Screening Visit or the participant has not stabilized from a previous relapse at the time of the Screening Visit.
* Current treatment with an investigational MS disease therapy.
* Prior treatment with:

Total lymphoid irradiation. Cladribine. T-cell or T-cell receptor vaccination. Campath-1h (alemtuzumab). Rituxan (rituximab).

* Prior treatment within three months with:

Tysabri (natalizumab). Gilenya (Fingolimod/FTY720). Zenapax (daclizumab). Cytoxan (cyclophosphamide). Novantrone (mitoxantrone). Cyclosporine. CellCept (mycophenolate mofetil). Imuran (azathioprine). Rheumatrex (methotrexate). IV gamma globulin. Plasma exchange.

* Prior treatment within one month:

Systemic corticosteroids with daily dose equivalent to Prednisone 60 mg or greater.

* Female participants who are not post-menopausal for at least one year, not surgically sterile, or not willing to practice effective contraception.
* Nursing mothers, pregnant women, or women planning to become pregnant during the study.
* Male participants who are not willing to practice effective contraception.
* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that, in the opinion of the Principal Investigator, is likely to affect the participant's ability to comply with the study protocol.
* Any other reason that, in the opinion of the Principal Investigator, makes the participant unsuitable for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of culturing MSCs, and infusion-related safety and tolerability of autologous MSC transplantation over one month in patients with relapsing forms of MS | 1 month

SECONDARY OUTCOMES:
To evaluate effects on MS disease activity measured by the number of Gd-enhancing brain MRI lesions | 1 month
To evaluate safety and tolerability of autologous MSC transplantation over 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Cohen, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Mellen Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Cohen JA, Imrey PB, Planchon SM, Bermel RA, Fisher E, Fox RJ, Bar-Or A, Sharp SL, Skaramagas TT, Jagodnik P, Karafa M, Morrison S, Reese Koc J, Gerson SL, Lazarus HM. Pilot trial of intravenous autologous culture-expanded mesenchymal stem cell transplantation in multiple sclerosis. Mult Scler. 2018 Apr;24(4):501-511. doi: 10.1177/1352458517703802. Epub 2017 Apr 6. PMID 28381130